CLINICAL TRIAL: NCT02612350
Title: Utility of Plasma Circulating Tumor DNA (ctDNA) in Asymptomatic Subjects for the Detection of Neoplastic Disease
Acronym: H1000
Status: Completed | Type: Observational
Sponsor: Pathway Genomics (Industry)
Responsible Party: Sponsor
Other Study IDs: Pathway Gennomics 004
Record Dates: First submitted 2015-11-13; First posted 2015-11-23 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Mutation; Neoplasms
Keywords: ctDNA; high risk for developing cancer; Plasma; Relative Risk; Early Detection of Cancer; Cancer Screening Tests; Cancer Screening
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be obtained, the plasma sample separated for the isolation of cell-free DNA, and the sample that may be stored will be excess plasma as well as potentially DNA from the buffy coat.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Increased Risk for Cancer Development: The group is to include at least 1000 individuals who are at high risk for the development of cancer. Risk is assessed through the completion of a clinical history questionnaire. Examples of such subjects include those with known hereditary cancer syndrome pathogenic variants without a diagnosis of cancer, with significant family history of breast, ovarian, colon, or lung cancer or melanoma, or another strong history of cancer but no prior molecular diagnosis, heavy smokers or those exposed to carcinogens and mutagens. The individuals who meet criteria for inclusion will undergo cell-free DNA isolation and circulating-tumor DNA (ctDNA) analysis for the detection of genetic mutations associated with the possible development of a malignancy.
  Interventions: Genetic: ctDNA Analysis for the Detection of Genetic Mutations

INTERVENTIONS:
Genetic: ctDNA Analysis for the Detection of Genetic Mutations — Cell-free DNA (cfDNA) is isolated from a blood plasma sample and tested for the presence of 96 specific well-described mutations in 9 cancer driver genes. The presence of more than 2 copies of a mutation may indicate the presence of a malignancy. Follow up with the subject's physician would be needed for an examination and any additional testing that the physician wants to perform to further assess for the development of cancer.

SUMMARY:
Pathway Genomics Corporation (Pathway Genomics), a San Diego, California company, is involved in the development and validation of new molecular diagnostic assays for the analysis of circulating tumor deoxyribonucleic acid (DNA) (ctDNA) found in the plasma-derived DNA (cell-free DNA or cfDNA) in order to identify specific variants (mutations) in cancer driver genes. The purpose of testing for mutations in ctDNA is to detect and monitor cancer. All cells shed DNA into the bloodstream. Finding cancer-associated mutations in the cfDNA may lead to early detection of cancer in an otherwise apparently healthy (i.e. asymptomatic) individual or may allow the healthcare provider to more effectively monitor and treat a known cancer patient. The analysis is performed using a polymerase chain reaction (PCR)-based methodology where oligonucleotides are designed to target specific mutations in designated genes of interest followed by next generation deep sequencing of the amplified targets. Evaluation of the performance of these assays for screening for cancer in asymptomatic subjects is essential for the clinical validation of the use of these assays. The specific aim of this protocol is to obtain relevant human blood samples from individual subjects at higher than average risk for the development of cancer due to age, heredity, or environmental or toxic exposures for use in the statistical analysis of this method as an adjunct screening test for the potential presence of cancer.

DETAILED DESCRIPTION:
The objectives of this study are to obtain human blood samples from asymptomatic subjects who have never been diagnosed with cancer, but who may be at increased risk for cancer due to heredity, exposures, age, or family history to assess the validity of screening healthy but at risk patients for cancer via analysis of ctDNA.

Specifically, the blood specimens will be collected from individuals who have responded to a self-administered health questionnaire that screens for higher risk of contracting cancer. Each participant will be asked to provide a 30 ml blood sample to be drawn by a primary care provider (PCP) or licensed phlebotomist. The specimens collected during the study may also be used in the research and development of new or modified molecular genetics assays. The results of these studies will be used to further the understanding of the use of ctDNA for the detection and monitoring of cancer in humans.

The blood samples are collected in blood collection tubes (BCT) called Cell-Free DNA BCT® manufactured by Streck and intended for collection, stabilization and transportation of cell-free plasma DNA. This device also stabilizes and preserves cellular genomic DNA present in nucleated blood cells and circulating epithelial cells (tumor cells) found in whole blood. This product has not been cleared by the U.S. Food and Drug Administration for In Vitro Diagnostic use and is labeled by Streck for research use only. Under the Clinical Laboratory Improvement Amendments (CLIA) regulations, laboratories are authorized to validate and use, as part of a laboratory-developed test (LDT), devices that have not been cleared or approved by the FDA. Pathway Genomics validated the CancerInterceptTM Detect molecular analysis system with the Streck tubes, in accordance with CLIA.

Once the specimen has been collected and sent to Pathway by the physician or the phlebotomist who collects the samples, all other processing and testing are conducted by Pathway laboratory personnel. The analysis begins with the separation of the plasma from the rest of the blood sample. cfDNA will then be isolated from each sample. The quantity of cfDNA is measured and then the sample is amplified via PCR for next generation sequencing. The results of the sequencing will then be analyzed for the presence of one or more of the 96 mutations analyzed in this assay. The data are then reviewed and a report will be generated.

ELIGIBILITY:
Inclusion Criteria:

* strong family history of cancer
* known carrier of a pathogenic variant in a gene indicating an increased risk of cancer, for example, in the BRCA1 or TP53 genes.
* exposure to environmental toxins, carcinogens, or mutagens, including but not limited to tobacco, radiation, asbestos, long-time industrial chemical exposure
* age equal to or over 50 years

Exclusion Criteria:

* prior diagnosis of cancer except basal cell carcinoma
* no risk factors that place the individual at high risk
* age under 18 years
* individuals unwilling to sign the IRB-approved consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are at increased risk for the development of cancer due to age over 50 years, a strong family history of cancer, known carrier of a pathogenic variant in a gene indicating an increased risk of cancer, for example a hereditary cancer syndrome, or due to exposure to environmental toxins, carcinogens, or mutagens, including tobacco. The individuals have to have the legal authority to provide consent, and therefore be 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 1106 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects found with one or more of 96 ctDNA mutations | 1 year
  A cohort of 1000 or more individuals who are at high risk for the development of cancer will be tested for the presence of 96 well-described mutations in 9 cancer driver genes via ctDNA analysis. The number of individuals with one or more of the 96 assayed mutations will be assessed.
Number of copies of mutant alleles found in the positive subjects | 1 year
  Among the cohort of subjects enrolled in the study in whom one or more of the 96 ctDNA mutations are detected, the number of copies per analyzed plasma sample will be calculated.
Percentage of ctDNA found within the total amount of circulating free DNA (cfDNA) | 1 year
  Within the samples found to contain one or more ctDNA mutation, the percentage of ctDNA within the total amount of cfDNA will be calculated.

SECONDARY OUTCOMES:
Number of subjects with one or more of 96 ctDNA mutations who develop cancer | 1 to 5 years
  The 1000 or more individuals in the study will be followed for 1 to 5 years to assess for the development of a malignancy. Special attention will be paid to the cohort who have initial assays indicating the presence of ctDNA. The subjects may be retested over time to show changing levels of ctDNA. Their own physicians will guide any follow up studies such as imaging or other laboratory testing. The test is designed as a means of case finding for cancer among individuals with high risk for development of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Braunstein, MD, Principal Investigator — Pathway Genomics; Anja Kammesheidt, PhD, Study Director — Pathway Genomics
Locations (1):
- Pathway Genomics, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidess E, Heirich K, Wiggin M, Vysotskaia V, Visser BC, Marziali A, Wiedenmann B, Norton JA, Lee M, Jeffrey SS, Poultsides GA. Mutation profiling of tumor DNA from plasma and tumor tissue of colorectal cancer patients with a novel, high-sensitivity multiplexed mutation detection platform. Oncotarget. 2015 Feb 10;6(4):2549-61. doi: 10.18632/oncotarget.3041. PMID 25575824
- [Background] Perrone F, Lampis A, Bertan C, Verderio P, Ciniselli CM, Pizzamiglio S, Frattini M, Nucifora M, Molinari F, Gallino G, Gariboldi M, Meroni E, Leo E, Pierotti MA, Pilotti S. Circulating free DNA in a screening program for early colorectal cancer detection. Tumori. 2014 Mar-Apr;100(2):115-21. doi: 10.1177/030089161410000201. PMID 24852853
- [Background] Lin PC, Lin JK, Lin CH, Lin HH, Yang SH, Jiang JK, Chen WS, Chou CC, Tsai SF, Chang SC. Clinical Relevance of Plasma DNA Methylation in Colorectal Cancer Patients Identified by Using a Genome-Wide High-Resolution Array. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S1419-27. doi: 10.1245/s10434-014-4277-2. Epub 2014 Dec 4. PMID 25472652
- [Background] Spindler KL, Appelt AL, Pallisgaard N, Andersen RF, Brandslund I, Jakobsen A. Cell-free DNA in healthy individuals, noncancerous disease and strong prognostic value in colorectal cancer. Int J Cancer. 2014 Dec 15;135(12):2984-91. doi: 10.1002/ijc.28946. Epub 2014 Jun 17. PMID 24798213
- [Background] Beaver JA, Jelovac D, Balukrishna S, Cochran R, Croessmann S, Zabransky DJ, Wong HY, Toro PV, Cidado J, Blair BG, Chu D, Burns T, Higgins MJ, Stearns V, Jacobs L, Habibi M, Lange J, Hurley PJ, Lauring J, VanDenBerg D, Kessler J, Jeter S, Samuels ML, Maar D, Cope L, Cimino-Mathews A, Argani P, Wolff AC, Park BH. Detection of cancer DNA in plasma of patients with early-stage breast cancer. Clin Cancer Res. 2014 May 15;20(10):2643-2650. doi: 10.1158/1078-0432.CCR-13-2933. Epub 2014 Feb 6. PMID 24504125
- [Background] Oshiro C, Kagara N, Naoi Y, Shimoda M, Shimomura A, Maruyama N, Shimazu K, Kim SJ, Noguchi S. PIK3CA mutations in serum DNA are predictive of recurrence in primary breast cancer patients. Breast Cancer Res Treat. 2015 Apr;150(2):299-307. doi: 10.1007/s10549-015-3322-6. Epub 2015 Mar 4. PMID 25736040
- [Background] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- [Background] Bianchi DW, Chudova D, Sehnert AJ, Bhatt S, Murray K, Prosen TL, Garber JE, Wilkins-Haug L, Vora NL, Warsof S, Goldberg J, Ziainia T, Halks-Miller M. Noninvasive Prenatal Testing and Incidental Detection of Occult Maternal Malignancies. JAMA. 2015 Jul 14;314(2):162-9. doi: 10.1001/jama.2015.7120. PMID 26168314
- [Background] Kinugasa H, Nouso K, Miyahara K, Morimoto Y, Dohi C, Tsutsumi K, Kato H, Matsubara T, Okada H, Yamamoto K. Detection of K-ras gene mutation by liquid biopsy in patients with pancreatic cancer. Cancer. 2015 Jul 1;121(13):2271-80. doi: 10.1002/cncr.29364. Epub 2015 Mar 30. PMID 25823825
- [Background] Sanmamed MF, Fernandez-Landazuri S, Rodriguez C, Zarate R, Lozano MD, Zubiri L, Perez-Gracia JL, Martin-Algarra S, Gonzalez A. Quantitative cell-free circulating BRAFV600E mutation analysis by use of droplet digital PCR in the follow-up of patients with melanoma being treated with BRAF inhibitors. Clin Chem. 2015 Jan;61(1):297-304. doi: 10.1373/clinchem.2014.230235. Epub 2014 Nov 19. PMID 25411185
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Hosny G, Farahat N, Tayel H, Hainaut P. Ser-249 TP53 and CTNNB1 mutations in circulating free DNA of Egyptian patients with hepatocellular carcinoma versus chronic liver diseases. Cancer Lett. 2008 Jun 18;264(2):201-8. doi: 10.1016/j.canlet.2008.01.031. Epub 2008 Mar 3. PMID 18313840
- [Background] Freidin MB, Freydina DV, Leung M, Montero Fernandez A, Nicholson AG, Lim E. Circulating tumor DNA outperforms circulating tumor cells for KRAS mutation detection in thoracic malignancies. Clin Chem. 2015 Oct;61(10):1299-304. doi: 10.1373/clinchem.2015.242453. Epub 2015 Aug 13. PMID 26272233
- [Background] Izumchenko E, Chang X, Brait M, Fertig E, Kagohara LT, Bedi A, Marchionni L, Agrawal N, Ravi R, Jones S, Hoque MO, Westra WH, Sidransky D. Targeted sequencing reveals clonal genetic changes in the progression of early lung neoplasms and paired circulating DNA. Nat Commun. 2015 Sep 16;6:8258. doi: 10.1038/ncomms9258. PMID 26374070
- [Background] Hamakawa T, Kukita Y, Kurokawa Y, Miyazaki Y, Takahashi T, Yamasaki M, Miyata H, Nakajima K, Taniguchi K, Takiguchi S, Mori M, Doki Y, Kato K. Monitoring gastric cancer progression with circulating tumour DNA. Br J Cancer. 2015 Jan 20;112(2):352-6. doi: 10.1038/bjc.2014.609. Epub 2014 Dec 9. PMID 25490524
- [Background] Wang Y, Springer S, Mulvey CL, Silliman N, Schaefer J, Sausen M, James N, Rettig EM, Guo T, Pickering CR, Bishop JA, Chung CH, Califano JA, Eisele DW, Fakhry C, Gourin CG, Ha PK, Kang H, Kiess A, Koch WM, Myers JN, Quon H, Richmon JD, Sidransky D, Tufano RP, Westra WH, Bettegowda C, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Agrawal N. Detection of somatic mutations and HPV in the saliva and plasma of patients with head and neck squamous cell carcinomas. Sci Transl Med. 2015 Jun 24;7(293):293ra104. doi: 10.1126/scitranslmed.aaa8507. PMID 26109104
- [Background] Reinert T, Scholer LV, Thomsen R, Tobiasen H, Vang S, Nordentoft I, Lamy P, Kannerup AS, Mortensen FV, Stribolt K, Hamilton-Dutoit S, Nielsen HJ, Laurberg S, Pallisgaard N, Pedersen JS, Orntoft TF, Andersen CL. Analysis of circulating tumour DNA to monitor disease burden following colorectal cancer surgery. Gut. 2016 Apr;65(4):625-34. doi: 10.1136/gutjnl-2014-308859. Epub 2015 Feb 4. PMID 25654990